CLINICAL TRIAL: NCT00345813
Title: Randomized Phase IIb Preprostatectomy Study of Dietary Supplementation With Soy and Biomarkers of Prostate Cancer Risk and Progression
Brief Title: Soy Supplements in Treating Patients Undergoing Surgery for Localized Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDR0000466317; CCCWFU-98203; CCCWFU-BG03-332
Record Dates: First submitted 2006-06-28; First posted 2006-06-29 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Soybean Proteins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (Experimental): Patients receive oral soy supplementation daily for 4 weeks. Patients undergo radical prostatectomy within 21 days after completion of soy supplementation.
  Interventions: Dietary Supplement: soy isoflavones; Dietary Supplement: soy protein isolate
- Arm II (Placebo Comparator): Patients receive oral placebo supplementation daily for 4 weeks. Patients undergo radical prostatectomy within 21 days after completion of placebo supplementation.
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: soy isoflavones — Given orally
  Arms: Arm I
Dietary Supplement: soy protein isolate — Given orally
  Arms: Arm I
Other: placebo — Given orally
  Arms: Arm II

SUMMARY:
RATIONALE: Dietary supplementation with soy may keep prostate cancer from growing in patients planning to undergo surgery.

PURPOSE: This randomized phase II trial is studying a soy supplement to see how well it works compared to a placebo in treating patients undergoing surgery for localized prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the effect of dietary supplementation with soy vs placebo on biomarkers of cell cycle regulation, proliferation, differentiation, apoptosis, and signaling pathways in patients with localized prostate cancer scheduled to undergo radical prostatectomy.

Secondary

* Compare the toxicity and side effects of these regimens in these patients.
* Compare the dietary patterns of these patients.

OUTLINE: This is a prospective, randomized study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral soy supplementation daily for 4 weeks.
* Arm II: Patients receive oral placebo supplementation daily for 4 weeks. Patients undergo radical prostatectomy within 21 days after completion of soy or placebo supplementation.

Blood and tissue samples are collected for biomarker analysis using immunohistochemistry.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * Clinically localized disease
* Scheduled for radical prostatectomy
* No evidence of metastatic disease by bone scan or CT scan of the abdomen or pelvis

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* No evidence of active nephrolithiasis
* No history of hypercalcemic syndrome

PRIOR CONCURRENT THERAPY:

* No prior treatment for prostate cancer, including radiotherapy, systemic chemotherapy, surgery, or investigational drugs
* No other concurrent dietary supplementation with soy, cholecalciferol (vitamin D), or fish oil

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2003-10; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Correlation of pretreatment ER-β expression with response to soy supplementation | within 21 days after completetion of supplement regimen
  after a 4 week therapy, within 21 days, a Radical Prostatectomy will be performed, and after that ER-β expression will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: M. Craig Hall, MD, Study Chair — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States